CLINICAL TRIAL: NCT04947436
Title: ALS and Airway Clearance (ALSAC) Is There a Best Therapy for Airway Clearance in Patients With ALS
Brief Title: ALS and Airway Clearance (ALSAC) Therapy
Acronym: ALSAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20120075
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Respiratory Muscle Weakness
Keywords: Amyotrophic Lateral Sclerosis; Airway Clearance; Mechanical Insufflation Exsufflation; High Frequency Chest Wall Compression Oscillation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Chest Wall Oscillation

STUDY DESIGN:
Intervention Model Description: A single-blind parallel group design in which 60 patients with probable or definite ALS will be randomized equally into three groups (20 per group) over a period of 12 months
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- High Frequency Chest Wall Oscillation (Active Comparator)
  Interventions: Device: High Frequency Chest Wall Oscillation
- Mechanical insufflation/ exsufflation (Active Comparator)
  Interventions: Device: Mechanical insufflation/exsufflation
- High Frequency Chest Wall Oscillation and Mechanical insufflation/ exsufflation (Active Comparator)
  Interventions: Device: High Frequency Chest Wall Oscillation; Device: Mechanical insufflation/exsufflation

INTERVENTIONS:
Device: High Frequency Chest Wall Oscillation — The HFCWO aims to mobilize the secretions to the pharynx to allow the patient to expel the secretions. However, many ALS patients are unable to expel their secretions due to atrophied expiratory muscles. The HFCWO device uses a small air compressor with a vest that wraps around the chest to induce airflows that pull secretions from the walls of the airways, thin the secretions and move them up the airways towards the larger airways and pharynx.
  Other Names: "The Vest"
  Arms: High Frequency Chest Wall Oscillation; High Frequency Chest Wall Oscillation and Mechanical insufflation/ exsufflation
Device: Mechanical insufflation/exsufflation — A noninvasive therapy, removes secretions in patients who have an ineffective cough because their peak cough flows are less than 270 L/min. This device applies a positive pressure to the airway and rapidly switches to a negative pressure applied to the airway. The rapid switch between the two types of pressure simulates a natural cough, thus assisting with expulsion of the secretions.
  Other Names: Cough Assist
  Arms: High Frequency Chest Wall Oscillation and Mechanical insufflation/ exsufflation; Mechanical insufflation/ exsufflation

SUMMARY:
Patients will receive one of three respiratory therapy interventions for airway clearance assistance: 1) High frequency chest wall oscillation (HFCWO) and mechanical insufflation/exsufflation (MIE), 2) HFCWO or 3) MIE. The study period will be six months and include three clinic visits, baseline and follow-up visits at 3 and 6 months, and 6 monthly home visits by the respiratory therapist.

DETAILED DESCRIPTION:
The proposed project includes both the HFCWO and MIE and will capitalize on the specific goals of each therapy and address the problem as a whole rather than piece-meal. The HFCWO aims to mobilize the secretions to the pharynx to allow the patient to expel the secretions. However, many patients diagnosed with ALS are unable to expel the secretions due to atrophied expiratory muscles. The HFCWO device uses a small air compressor with a vest that wraps around the chest to induce airflows to pull secretions from the walls of the airways, thin the secretions and move them up the airways towards the larger airways and pharynx. The MIE, a noninvasive therapy, removes secretions in patients who have an ineffective cough because the peak cough flows are less than 270 L/min. This device applies a positive pressure to the airway and rapidly switches to a negative pressure applied to the airway. The rapid switch between the two types of pressure simulates a natural cough, thus assisting with expulsion of the secretions. Logically, the two mechanisms of action of these devices should work synergistically to produce effective airway clearance to keep the lungs clear, healthy and reduce the risk of infections from stagnant secretions. Respiratory infections are especially serious for patients with ALS because the patient is not able to recuperate from infections as quickly as a person without ALS. The objective is to determine if changing the use of existing respiratory therapy devices can improve the physical and psychosocial health and quality of life for patients diagnosed with ALS and caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 and above,
2. Probable or definite ALS diagnosis,
3. Peak Cough Flow of <160L/min or complain of issues clearing airway secretions
4. Caregiver must also consent to participate

Exclusion Criteria:

1. Current use of HFCWO or MIE
2. Tracheostomy
3. Congestive heart failure
4. All contraindications for the HFCWO
5. Head and/or neck injury that has not been stabilized;
6. Active hemorrhage with hemodynamic instability;
7. Uncontrolled hypertension;
8. Active or recent gross hemoptysis; and
9. All contraindications for the MIE
10. History of bullous emphysema;
11. Known susceptibility to pneumothorax;
12. Pneumomediastinum; and
13. Recent barotrauma
14. Frontal Temporal Dementia (FTD) - suspected or diagnosed . FTD is a form of dementia found in about 20% of Familial ALS. This dementia interferes with the ability to follow commands and follow through with therapies due to forgetfulness.
15. Patients not able to provide informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2017-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Gardner, DrPH, Principal Investigator — University of Texas Health San Antonio
Locations (1):
- University of Texas Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be available in result publication and in summary result reporting in ClinicalTrials.gov
Supporting Information: SAP
Time Frame: In a peer review journal post study completion and data analysis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients and their caregivers (PAC) were randomized into one of three groups. The PAC completed perception of problem and quality of life surveys.
Period: Overall Study
Arm/Group | High Frequency Chest Wall Oscillation | Mechanical Insufflation/ Exsufflation | High Frequency Chest Wall Oscillation and Mechanical Insufflation/ Exsufflation
Started | 7 | 10 | 11
Completed | 3 | 2 | 5
Not Completed | 4 | 8 | 6
Not completed — Lost to Follow-up | 3 | 7 | 5
Not completed — Death | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Frequency Chest Wall Oscillation | High Frequency Chest Wall Oscillation and Mechanical Insufflation/ Exsufflation | Mechanical Insufflation/ Exsufflation | Total
Number analyzed (Participants) | 7.0 | 11.0 | 10.0 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 3 | 14
  >=65 years | 3 | 4 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 3 | 7 | 5 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic-Non White | 2 | 3 | 2 | 7
  White | 5 | 6 | 7 | 18
  Black | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Complications Severity
Description: A 9-item instrument will be used to record change from baseline to 6 months in respiratory complications. These are scored on a scale from best (no complications) to worst (death due to respiratory complications) throughout the study period. Scores range from 0-9 with a score of a 9 indicating no complications.
Time Frame: Baseline to 6 months
Population: Half (50%) of patients were randomized to the group with two devices, while 30% to only the HFCWO device and 20% to only the Mechanical Insufflation/exsufflation device.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Chest Wall Oscillation | Mechanical Insufflation/ Exsufflation | High Frequency Chest Wall Oscillation and Mechanical Insufflation/ Exsufflation
Number analyzed (Participants) | 3 | 2 | 5
score on a scale | 8.33 (1.15) | 9.0 (0) | 7.8 (1.64)

2. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: This outcome is assessed and recorded as a number from 1-5 with 1 indicating the worst outcome (markedly worse) and 5 indicating best outcome (markedly better) since starting the study.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Chest Wall Oscillation | Mechanical Insufflation/ Exsufflation | High Frequency Chest Wall Oscillation and Mechanical Insufflation/ Exsufflation
Number analyzed (Participants) | 3 | 2 | 5
score on a scale | 3.33 (0.58) | 3.00 (0) | 4.40 (0.96)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All adverse events were collected during participant enrollment period in the study, regardless of whether or not they were related to treatment or condition.
Arm/Group | High Frequency Chest Wall Oscillation | Mechanical Insufflation/ Exsufflation | High Frequency Chest Wall Oscillation and Mechanical Insufflation/ Exsufflation
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/10 | 1/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
Limitations include small sample size due to length of time associated with the intervention and the progression of the disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes